CLINICAL TRIAL: NCT00616707
Title: Analysis of Microalbuminuria and Markers of Inflammation and Oxidative Stress in Adolescents of Different Ethnic Backgrounds
Acronym: IM
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Sponsor
Other Study IDs: 200614513
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Inflammation
Keywords: Inflammation; Oxidative Stress; Microalbuminuria
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Aliquots from the citrate vial & Serum seperator vial are being retained
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if there are signs of inflammation in one's blood and urine and to find out if one's body size or ethnicity has an effect on these substances.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 12 to 18 years old
* Hispanic, African American or Caucasian ethnicity
* Have a Body Mass Index (BMI) between the 5th and 85th percentile or greater than the 95th percentile
* Must currently be attending a UC Davis Pediatric clinic

Exclusion Criteria:

* Chronic liver or kidney disease, known Diabetes or other chronic illnesses (such as Sickle Cell Disease or Cystic Fibrosis)
* Subjects can NOT be acutely febrile, smoke, chronically use prescription medications or oral contraceptive pills.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric out-patient at UCDavis Medical Center clinic
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2006-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To compare plasma levels of inflammatory markers and urinary biomarkers of oxidative stress in adolescents of Hispanic, African-American and Caucasian ethnicity | at the end of study

SECONDARY OUTCOMES:
To determine if there is an independent correlation between these markers and urinary microalbumin excretion | at the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Lavjay Butani, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- See also: Related Info — http://www.ucdmc.ucdavis.edu/clinicaltrials/trialDetail.aspx?protocol=200614513